CLINICAL TRIAL: NCT03689582
Title: 68GA-PSMA Fusion PET/MRI For Image-Guided Prostate Biopsies
Brief Title: Radiolabeled Gallium-68 (68Ga-PSMA) for PET/CT Imaging to Detect Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to pandemic related constraints
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UMCC 2018.072; HUM00146602 (Other: University of Michigan)
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Results first posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA (Experimental): PET/CT imaging with 68Ga-PSMA
  Interventions: Drug: 68Ga-PSMA

INTERVENTIONS:
Drug: 68Ga-PSMA — Positron Emission Tomography/Computed Tomography (PET/CT) imaging with 68Ga-PSMA:
  68Ga-PSMA is an investigational radioactive drug that binds to receptors on prostate cancer cells. The intravenously administered drug dose will be about 5 mCi (range 3-7 mCi).
  Other Names: Gallium-68 PSMA-HBED-CC; Gallium-68 PSMA-11

SUMMARY:
The purpose of the study is to find out whether imaging of the prostate with a new molecule called 68Ga-PSMA can find prostate cancer. 68Ga-PSMA has been shown in a large number of patients to be useful to find recurring prostate cancer following initial cancer treatment. This study is performed to test 68Ga-PSMA whether it can be used to find prostate cancers that would be considered in need for treatment.

DETAILED DESCRIPTION:
In this study, two different imaging tests are being compared: a) 68Ga-PSMA Positron Emission Tomography (PET)/Computed Tomography (CT) and b) Magnetic Resonance Imaging (MRI) of the prostate gland. Participants already have received the MRI, and the results were either suspicious of or definitive for prostate cancer. Both tests (MRI and 68Ga-PSMA PET/CT) are expected to show tumor tissue when more aggressive, but one test could be more accurate than the other test.

Another important question is whether these imaging tests will perform as good or better than prostate biopsies in finding all prostate cancer lesions in need for treatment. If imaging would be comparable or better than biopsies, then imaging may be able to replace invasive biopsies for some indications in the future.

To investigate these questions, participants are asked to undergo a 68Ga-PSMA PET/CT before a planned prostate biopsy procedure. After the biopsy procedure is performed, investigators will compare the imaging results from 68Ga-PSMA with those from the MRI and determine which test is more accurate.

ELIGIBILITY:
Inclusion Criteria:

* Recent MRI of the prostate has resulted in at least one lesion suspected to represent prostate cancer (reported by the Radiologist as PI-RADS 3, 4 or 5 lesion)
* Treating physician has already indicated a need for a prostate biopsy procedure.
* Known Gleason 6 or 7 prostate cancer OR rising PSA with either a) no prior biopsy or b) single or multiple negative prior biopsies.

Exclusion Criteria:

* Prostate biopsy within 12 weeks before enrollment
* Acute prostatitis within the last 6 months
* Current non-urologic bacterial infection requiring active treatment with antibiotics
* Active other malignancy (except basal cell or squamous cell skin cancer) within the last 2 years
* Body weight greater than 350 lbs (158 Kg)
* Inability or unwillingness to receive a prostate biopsy procedure
* Unable to lie flat, still, or tolerate a PET/CT scan
* Unable to provide own consent
* Concurrent severe and/or uncontrolled and/or unstable medical disease other than prostate cancer (e.g. poorly controlled diabetes, congestive heart failure, myocardial infarction within 6 months prior to study participation, unstable and uncontrolled hypertension, acute renal failure of any intensity, chronic renal or hepatic disease, severe pulmonary disease).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morand R Piert, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Codified data will be archived and stored in an imaging repository with limited metadata for analysis. Individuals seeking use of these data should contact the study chair. A data sharing contract for a HIPAA limited dataset will need to be executed prior to data sharing.
Supporting Information: CSR
Time Frame: Available as requested. Data will be archived indefinitely for research purposes.
Access Criteria: Individuals seeking use of these data should contact the study chair.

REFERENCES:
- [Background] Hicks RM, Simko JP, Westphalen AC, Nguyen HG, Greene KL, Zhang L, Carroll PR, Hope TA. Diagnostic Accuracy of 68Ga-PSMA-11 PET/MRI Compared with Multiparametric MRI in the Detection of Prostate Cancer. Radiology. 2018 Dec;289(3):730-737. doi: 10.1148/radiol.2018180788. Epub 2018 Sep 18. PMID 30226456

RESULTS

PARTICIPANT FLOW:
Groups:
- 68Ga-PSMA: PET/CT imaging with 68Ga-PSMA: 68Ga-PSMA is an investigational radioactive drug that binds to receptors on prostate cancer cells. The intravenously administered drug dose will be about 5 mCi (range 3-7 mCi).
Period: Overall Study
Arm/Group | 68Ga-PSMA
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 68Ga-PSMA
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 71 [53 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Two Different Radiologic Imaging Techniques, Fusion PET/MRI and Standard MRI, With Histopathologic Reference Data From Prostate Biopsy
Description: Fusion PET/MRI is the combination of 68Ga-PSMA Positron Emission Tomography/Computed Tomography (PET/CT) plus Multiparametric MRI (mpMRI)-guided biopsy. Reference standard will be pathology-defined as targeted plus standard prostate biopsy, and prostatectomy, when available. The original intent was to determine the sensitivity and specificity of standard-of-care Multiparametric MRI (mpMRI) alone (using PI-RADS version 2) and fusion PET/MRI for the detection of primary Gleason ≥3+4 cancer, and to estimate the positive likelihood ratio (LR) of each. However, due to pandemic-related early closure of the study, enrollment was less than 15% of the enrolment goal necessary to achieve statistical power. Therefore, it is not possible to responsibly report the originally listed outcome measure of likelihood ratio. Instead, the results table displays the summary of collected imaging data, categorized by type of scan, in comparison to the reference standard histopathology.
Time Frame: Up to ~4 weeks (after planned, standard-of-care biopsy).
Measure: Number; unit: participants
Groups:
- Histology Result of Biopsy: Prostate Cancer: Participants whose histology result of biopsy is prostate cancer.
- Benign Histology Result: Participants whose histology result of biopsy is benign.
Arm/Group | Histology Result of Biopsy: Prostate Cancer | Benign Histology Result
Number analyzed (Participants) | 11 | 11
participants
  PSMA scan true positive and MRI scan true positive | 7 | 0
  PSMA scan true positive and MRI scan false negative | 2 | 0
  PSMA scan false negative and MRI scan false negative | 1 | 0
  PSMA scan true negative and MRI scan true negative | 0 | 1

2. Secondary Outcome: Adverse Events of 68Ga-PSMA Administration
Description: Adverse events will be determined through clinical assessment and categorized by CTCAE 4.0.
Time Frame: 24 hours post injection
Measure: Number; unit: adverse events
Arm/Group | 68Ga-PSMA
Number analyzed (Participants) | 11
adverse events | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | 68Ga-PSMA
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 68Ga-PSMA (N=11)
Claustrophobia (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT03689582/Prot_SAP_000.pdf